CLINICAL TRIAL: NCT03808272
Title: A Prospective, Multi-center, Single-arm Study to Evaluate the Safety and Efficacy of AXIOS Stent and Electrocautery-enhanced Delivery System in Chinese Patients With Pancreatic Pseudocyst and Walled-off Necrosis(WON)
Brief Title: AXIOS CHINA (E7148)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7148
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Pseudocyst and Walled-off Necrosis
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HOT AXIOS Stent and Electrocautery- Enhanced Delivery System (Experimental): HOT AXIOS Stent and Electrocautery- Enhanced Delivery System
  Interventions: Device: HOT AXIOS Stent and Electrocautery- Enhanced Delivery System

INTERVENTIONS:
Device: HOT AXIOS Stent and Electrocautery- Enhanced Delivery System — The HOT AXIOS Stent and Electrocautery- Enhanced Delivery System is indicated for use to facilitate transgastric or transduodenal endoscopic drainage of a pancreatic pseudocyst or a walled-off necrosis with ≥ 70% fluid content.

SUMMARY:
To study the safety and effectiveness of the AXIOS Stent with Electrocautery Enhanced Delivery System for endoscopic trans enteric drainage of pancreatic pseudocyst and walled-off necrosis in Chinese population, to support the regulatory approval by CFDA

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old(including 18 and 75 years old)
2. Eligible for endoscopic intervention
3. Acceptable candidate for endoscopic transluminal pancreatic pseudocyst drainage
4. Diagnostic as symptomatic pancreatic pseudocysts ≥ 6cm in maximum diameter and walled-off necrosis ≥ 6cm in maximum diameter with ≥ 70% fluid content that are adherent to the gastric or bowel wall
5. Patient understands the study requirements and the treatment procedures and provides written Informed Consent.
6. Patient is willing to comply with all specified follow-up evaluations, including willingness to undergo a pre/post CT imaging study.

Exclusion Criteria:

1. <18 or >75 years of age
2. pseudocysts or walled-off necrosis which require nasocystic drainage,or<6cm in maximum diameter, or walled-off necrosis < 70% fluid content
3. The fluid collection to be drained is an immature pseudocyst
4. The fluid collection to be drained is a cystic neoplasm
5. The fluid collection to be drained is a pseudoaneurysm
6. The fluid collection to be drained is a duplication cyst
7. The fluid collection to be drained is a non-inflammatory fluid collection
8. There is more than one pseudocyst requiring drainage
9. Abnormal coagulation: INR > 1.5 and not correctable presence of a bleeding disorder; platelets < 50,000/mm3
10. Altered anatomy that precludes the physician's ability to deliver the stent (decision on a case by case basis).
11. Intervening gastric varices or vessels within a one centimeter radius of the needle (visible using endoscopy or endoscopic ultrasound)
12. Any prior true anaphylactic reaction to contrast agents, nitinol (nickel titanium), silicone or any other materials contacting the patient.
13. Female of childbearing potential with a positive pregnancy test prior to the procedure or intends to become pregnant during the study.
14. Currently participating in another investigational drug of device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Technical success rate | 28± 7 days post stent placement
  defined as: placement of the AXIOS stent using the Electrocautery Enhanced AXIOS delivery system and removal of the AXIOS stent using a standard method: such as endoscopic snare or forceps.
Clinical success rate | 28± 7 days post stent placement
  defined as: at least a 50% decrease in pseudocyst's maximum diameter, based on radiographic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Shutian Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No